CLINICAL TRIAL: NCT02494583
Title: A Randomized, Active-Controlled, Partially Blinded, Biomarker Select, Phase III Clinical Trial of Pembrolizumab as Monotherapy and in Combination With Cisplatin+5-Fluorouracil Versus Placebo+Cisplatin+5-Fluorouracil as First-Line Treatment in Subjects With Advanced Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Study of Pembrolizumab (MK-3475) as First-Line Monotherapy and Combination Therapy for Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (MK-3475-062/KEYNOTE-062)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-062; 163187 (Registry Identifier: JAPIC-CTI); MK-3475-062 (Other: Merck Protocol Number); KEYNOTE-062 (Other: Merck); 2015-000972-88 (EudraCT Number)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Results first posted 2020-03-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric carcinoma; Gastric cancer; Gastroesophageal junction cancer; Gastroesophageal junction carcinoma; Programmed Cell Death-1 (PD1, PD-1),; Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Fluorouracil; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is partially blinded. The participant, study site personnel, and the sponsor will be blinded in the pembrolizumab plus SOC chemotherapy (pembro combo) arm and the placebo plus SOC chemotherapy (SOC) arm, but not in the pembro monotherapy (mono arm) since only one type of study medication will be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab Monotherapy (Pembro Mono) (Experimental): Participants will receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W). Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab + SOC Chemotherapy (Pembro Combo) (Experimental): Participants will receive pembrolizumab 200 mg Q3W plus cisplatin 80 mg/m^2 Q3W plus 5-FU 800 mg/m^2/day IV infusion on Days 1-5 Q3W. Capecitabine 1000 mg/m^2 twice a day (BID) on Days 1-14 Q3W may be substituted for 5-FU per local guidelines. Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: 5-FU; Drug: Capecitabine
- Placebo + SOC Chemotherapy (SOC) (Placebo Comparator): Participants receive placebo IV Q3W plus cisplatin 80 mg/m^2 Q3W plus 5-FU 800 mg/m^2/day IV infusion on Days 1-5 Q3W. Capecitabine 1000 mg/m^2 BID on Days 1-14 Q3W may be substituted for 5-FU per local guidelines.
  Interventions: Drug: Cisplatin; Drug: 5-FU; Drug: Capecitabine; Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab 200 mg IV on Day 1 of each week in 3-week cycles for up to 35 cycles (approximately 2 years).
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + SOC Chemotherapy (Pembro Combo); Pembrolizumab Monotherapy (Pembro Mono)
Drug: Cisplatin — Cisplatin 80 mg/m^2 IV on Day 1 of each week in 3-week cycles (6 cycle maximum per local country guidelines).
  Arms: Pembrolizumab + SOC Chemotherapy (Pembro Combo); Placebo + SOC Chemotherapy (SOC)
Drug: 5-FU — 5-FU 800 mg/m^2/day IV continuous from Day 1-5 of each 3-week cycle.
  Arms: Pembrolizumab + SOC Chemotherapy (Pembro Combo); Placebo + SOC Chemotherapy (SOC)
Drug: Capecitabine — Capecitabine 1000 mg/m^2 twice daily by oral tablet on Day 1-14 of each 3-week cycle.
  Arms: Pembrolizumab + SOC Chemotherapy (Pembro Combo); Placebo + SOC Chemotherapy (SOC)
Drug: Placebo — Normal saline IV on Day 1 of each week in 3-week cycles for up to 35 cycles (approximately 2 years).
  Arms: Placebo + SOC Chemotherapy (SOC)

SUMMARY:
This is a study of pembrolizumab (MK-3475) as first-line treatment for participants with advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma. Participants whose tumors express programmed death-ligand 1 (PD-L1) will be randomly assigned to one of the three treatment arms of the study: pembrolizumab as monotherapy [pembro mono], pembrolizumab plus standard of care (SOC) chemotherapy with cisplatin plus 5-fluorouracil (5-FU) or capecitabine [pembro combo], or placebo plus SOC chemotherapy with cisplatin plus 5-fluorouracil (5-FU) or capecitabine [SOC].

The primary study hypotheses are that pembrolizumab in combination with SOC chemotherapy is superior to SOC chemotherapy alone in terms of Progression-free Survival (PFS) and Overall Survival (OS) in participants with PD-L1 Combined Positive Score (CPS) ≥1, pembrolizumab in combination with SOC chemotherapy is superior to SOC chemotherapy alone in terms of OS in participants with PD-L1 CPS ≥10, pembrolizumab monotherapy is non-inferior to SOC chemotherapy alone in terms of OS in participants with PD-L1 CPS ≥1, and pembrolizumab monotherapy is superior to SOC chemotherapy alone in terms of OS in participants with PD-L1 CPS ≥1 and in participants with PD-L1 CPS ≥10.

DETAILED DESCRIPTION:
As specified by the protocol, primary and secondary efficacy analyses will be evaluated in gastric cancer participants with PD-L1 CPS ≥1 (all participants) and PD-L1 CPS ≥10 (OS) by comparing the pembro mono arm or pembro combo arm separately to the SOC arm.

ELIGIBILITY:
Inclusion Criteria:

* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 3 days prior to first dose of study medication
* Has histologically- or cytologically-confirmed diagnosis of locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma
* Human epidermal growth factor receptor 2- (HER2/neu-) negative and programmed cell death ligand 1 (PD-L1)-positive
* Has measurable disease
* Female participants of childbearing potential must be willing to use adequate contraception or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
* Male participants of childbearing potential should agree to use an adequate method of contraception starting with the first dose of study medication through 120 days after the last dose of study medication
* Adequate organ function

Exclusion Criteria:

* Squamous cell or undifferentiated gastric cancer
* Previous therapy for locally advanced, unresectable or metastatic gastric/GEJ cancer. Participant may have received prior neoadjuvant or adjuvant therapy as long as it was completed at least 6 months prior to randomization
* Major surgery, open biopsy or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of study treatment.
* Radiotherapy within 14 days of randomization
* Known additional malignancy that is progressing or requires active treatment with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in past 2 years
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* History of non-infectious pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of study medication
* Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, or anti-PD-L2 agent
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or C
* Currently participating in and receiving study therapy or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study medication
* Received a live vaccine within 30 days prior to the first dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Janjigian YY, Cecchini M, Shitara K, Enzinger PC, Wainberg ZA, Chau I, Satoh T, Lee J, Nebozhyn M, Loboda A, Kobie J, Vajdi A, Shih CS, Cristescu R, Cao ZA. Genomic Landscape of Late-Stage Gastric Cancer: Analysis From KEYNOTE-059, KEYNOTE-061, and KEYNOTE-062 Studies. JCO Precis Oncol. 2025 Mar;9:e2400456. doi: 10.1200/PO-24-00456. Epub 2025 Mar 21. PMID 40117530
- [Derived] Muro K, Shitara K, Yamaguchi K, Yoshikawa T, Satake H, Hara H, Sugimoto N, Machida N, Goto M, Kawakami H, Amagai K, Omuro Y, Esaki T, Hironaka S, Nishina T, Komatsu Y, Matsubara H, Shiratori S, Han S, Satoh T, Ohtsu A. Efficacy of Pembrolizumab Monotherapy in Japanese Patients with Advanced Gastric or Gastroesophageal Junction Cancer. J Gastrointest Cancer. 2023 Sep;54(3):951-961. doi: 10.1007/s12029-023-00920-9. Epub 2023 Apr 10. PMID 37037952
- [Derived] Satake H, Lee KW, Chung HC, Lee J, Yamaguchi K, Chen JS, Yoshikawa T, Amagai K, Yeh KH, Goto M, Chao Y, Lam KO, Han SR, Shiratori S, Shah S, Shitara K. Pembrolizumab or pembrolizumab plus chemotherapy versus standard of care chemotherapy in patients with advanced gastric or gastroesophageal junction adenocarcinoma: Asian subgroup analysis of KEYNOTE-062. Jpn J Clin Oncol. 2023 Mar 7;53(3):221-229. doi: 10.1093/jjco/hyac188. PMID 36533429
- [Derived] Lee KW, Van Cutsem E, Bang YJ, Fuchs CS, Kudaba I, Garrido M, Chung HC, Lee J, Castro HR, Chao J, Wainberg ZA, Cao ZA, Aurora-Garg D, Kobie J, Cristescu R, Bhagia P, Shah S, Tabernero J, Shitara K, Wyrwicz L. Association of Tumor Mutational Burden with Efficacy of Pembrolizumab+/-Chemotherapy as First-Line Therapy for Gastric Cancer in the Phase III KEYNOTE-062 Study. Clin Cancer Res. 2022 Aug 15;28(16):3489-3498. doi: 10.1158/1078-0432.CCR-22-0121. PMID 35657979
- [Derived] Chao J, Fuchs CS, Shitara K, Tabernero J, Muro K, Van Cutsem E, Bang YJ, De Vita F, Landers G, Yen CJ, Chau I, Elme A, Lee J, Ozguroglu M, Catenacci D, Yoon HH, Chen E, Adelberg D, Shih CS, Shah S, Bhagia P, Wainberg ZA. Assessment of Pembrolizumab Therapy for the Treatment of Microsatellite Instability-High Gastric or Gastroesophageal Junction Cancer Among Patients in the KEYNOTE-059, KEYNOTE-061, and KEYNOTE-062 Clinical Trials. JAMA Oncol. 2021 Jun 1;7(6):895-902. doi: 10.1001/jamaoncol.2021.0275. PMID 33792646
- [Derived] Shitara K, Van Cutsem E, Bang YJ, Fuchs C, Wyrwicz L, Lee KW, Kudaba I, Garrido M, Chung HC, Lee J, Castro HR, Mansoor W, Braghiroli MI, Karaseva N, Caglevic C, Villanueva L, Goekkurt E, Satake H, Enzinger P, Alsina M, Benson A, Chao J, Ko AH, Wainberg ZA, Kher U, Shah S, Kang SP, Tabernero J. Efficacy and Safety of Pembrolizumab or Pembrolizumab Plus Chemotherapy vs Chemotherapy Alone for Patients With First-line, Advanced Gastric Cancer: The KEYNOTE-062 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1571-1580. doi: 10.1001/jamaoncol.2020.3370. PMID 32880601
- See also: Merck Oncology Clinical Trial Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma who were programmed death-ligand 1 (PD-L1)-positive (Combined Positive Score [CPS]≥1) and human epidermal growth factor receptor 2 (HER2/neu)-negative were recruited to the study.
Pre-assignment Details: Of 1,787 screened, 763 were randomized 1:1:1 to the pembrolizumab monotherapy (pembro mono) arm, pembrolizumab plus standard of care (SOC) chemotherapy (pembro combo) arm, or placebo plus SOC chemotherapy (SOC) arm. Per protocol, response/progression or adverse events (AEs) that occurred during the second course were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Pembrolizumab Monotherapy (Pembro Mono): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W). Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Pembrolizumab + SOC Chemotherapy (Pembro Combo): Participants received pembrolizumab 200 mg Q3W plus cisplatin 80 mg/m^2 Q3W plus 5-fluorouracil (5-FU) 800 mg/m^2/day IV infusion on Days 1-5 Q3W. Capecitabine 1000 mg/m^2 twice a day (BID) on Days 1-14 Q3W could be substituted for 5-FU per local guidelines. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Placebo + SOC Chemotherapy (SOC): Participants received placebo IV Q3W plus cisplatin 80 mg/m^2 Q3W plus 5-FU 800 mg/m^2/day IV infusion on Days 1-5 Q3W. Capecitabine 1000 mg/m^2 BID on Days 1-14 Q3W could be substituted for 5-FU per local guidelines.
Period: Overall Study
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Started | 256 | 257 | 250
Received First Course of Pembrolizumab | 254 (1 participant randomized to the pembro combo arm received pembrolizumab monotherapy by mistake.) | 250 | 244
Received Second Course of Pembrolizumab | 4 | 5 | 0
Completed | 0 | 0 | 0
Not Completed | 256 | 257 | 250
Not completed — Death | 224 | 214 | 225
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Screen Failure | 0 | 1 | 0
Not completed — Transferred to Extension Study | 15 | 15 | 6
Not completed — Did Not Continue on Extension Study | 8 | 10 | 4
Not completed — Withdrawal by Subject | 7 | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC) | Total
Number analyzed (Participants) | 256 | 257 | 250 | 763
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (11.6) | 60.9 (11.6) | 60.7 (12.7) | 60.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 62 | 71 | 209
  Male | 180 | 195 | 179 | 554
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 54 | 46 | 145
  Not Hispanic or Latino | 206 | 196 | 197 | 599
  Unknown or Not Reported | 5 | 7 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 7 | 13 | 29
  Asian | 69 | 71 | 67 | 207
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 4 | 4 | 5 | 13
  White | 164 | 167 | 154 | 485
  More than one race | 9 | 6 | 7 | 22
  Unknown or Not Reported | 0 | 2 | 3 | 5
Region of Enrollment [Number; unit: Participants] — Participants were stratified according to geographic region of enrolling site:
  Europe (including Israel)/North America/Australia, Asia (including East Asia [South Korea, Hong Kong, Taiwan], South East Asia [Malaysia], Thailand, Singapore, Japan), or Rest of the World (including South America).
  Participants
    Europe/North America/Australia | 148 | 148 | 147 | 443
    Asia | 62 | 64 | 61 | 187
    Rest of the World | 46 | 45 | 42 | 133
Disease Status [Count of Participants; unit: Participants] — Participants were stratified according to gastric cancer disease status as either locally advanced unresectable or metastatic disease.
  Participants
    Locally advanced | 10 | 12 | 13 | 35
    Metastatic | 245 | 243 | 235 | 723
    Missing | 1 | 2 | 2 | 5
Fluoropyrimidine Treatment [Count of Participants; unit: Participants] — Participants receiving SOC chemotherapy were stratified according to fluoropyrimidine treatment (5-FU or capecitabine).
  Participants
    5-FU | 97 | 98 | 95 | 290
    Capecitabine | 159 | 159 | 155 | 473

OUTCOME MEASURES:

1. Primary Outcome: Pembro Combo vs SOC: Progression Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) in Participants With PD-L1 CPS ≥1 (All Participants)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro combo arm was compared to the SOC arm as a pre-specified primary analysis of the Intent-To-Treat (ITT) population. PFS is reported here for all participants in the pembro combo arm and SOC arm who were PD-L1 CPS ≥1 (all participants). Per protocol, PFS was compared separately between CPS ≥1 participants of the pembro mono arm and SOC arm and is presented later in the record.
Time Frame: Up to approximately 36 months
Population: All CPS ≥1 participants in the ITT population randomized to the pembro combo arm and SOC arm were analyzed. Per protocol, the pembro mono arm was compared to the SOC arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab Monotherapy (Pembro Mono): Participants received pembrolizumab 200 mg IV Q3W.
- Pembrolizumab + SOC Chemotherapy (Pembro Combo): Participants received pembrolizumab 200 mg Q3W plus cisplatin 80 mg/m^2 Q3W plus 5-FU 800 mg/m^2/day IV infusion on Days 1-5 Q3W. Capecitabine 1000 mg/m^2 twice a day (BID) on Days 1-14 Q3W could be substituted for 5-FU per local guidelines.
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 0 | 257 | 250
Months |  | 6.9 [5.7 to 7.3] | 6.4 [5.7 to 7.0]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC Chemotherapy (Pembro Combo) vs Placebo + SOC Chemotherapy (SOC); PFS in CPS ≥1 participants of the pembro combo arm was compared to PFS in CPS ≥1 participants of the SOC arm to address the first primary hypothesis (superiority to SOC). The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification according to geographic region, disease status, and fluoropyrimidine treatment; Test type: Superiority; p = 0.03918, Regression, Cox — One-sided p-value based on log-rank test with stratification; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.70 to 1.02] — Since stratified analyses could be based on collapsing strata with insufficient number of participants or events, strata were pooled in some cases based on clinical judgement and actual counts

2. Primary Outcome: Pembro Combo vs SOC: Overall Survival (OS) in Participants With PD-L1 CPS ≥1 (All Participants)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro combo arm was compared to the SOC arm as a pre-specified primary analysis of the ITT population. OS is reported here for all participants in the pembro combo arm and SOC arm who were PD-L1 CPS ≥1 (all participants). Per protocol, OS was compared separately between CPS ≥1 participants of the pembro mono arm and SOC arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 0 | 257 | 250
Months |  | 12.5 [10.8 to 13.9] | 11.1 [9.2 to 12.8]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC Chemotherapy (Pembro Combo) vs Placebo + SOC Chemotherapy (SOC); OS in CPS ≥1 participants of the pembro combo arm was compared to OS in CPS ≥1 participants of the SOC arm to address the second primary hypothesis (superiority to SOC). The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification according to geographic region, disease status, and Fluoropyrimidine treatment; Test type: Superiority; p = 0.04611, Regression, Cox — One-sided p-value based on log-rank test with stratification; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.03] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Pembro Combo vs SOC: OS in Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro combo arm was compared to the SOC arm as a pre-specified primary analysis of the ITT population. OS is reported here for all participants in the pembro combo arm and SOC arm who were PD-L1 CPS ≥10. Per protocol, OS was compared separately between CPS ≥10 participants of the pembro mono arm and SOC arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: All CPS ≥10 participants in the ITT population randomized to the pembro combo arm and SOC arm were analyzed. Per protocol, the pembro mono arm was compared to the SOC arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 0 | 99 | 90
Months |  | 12.3 [9.5 to 14.8] | 10.8 [8.5 to 13.8]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC Chemotherapy (Pembro Combo) vs Placebo + SOC Chemotherapy (SOC); OS in CPS ≥10 participants of the pembro combo arm was compared to OS in CPS ≥10 participants of the SOC arm to address the third primary hypothesis (superiority to SOC). The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification according to geographic region, disease status, and Fluoropyrimidine treatment; Test type: Superiority; p = 0.15804, Regression, Cox — One-sided p-value based on log-rank test with stratification; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.62 to 1.17] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Pembro Mono vs SOC: OS in Participants With PD-L1 CPS ≥1 (All Participants)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro mono arm was compared to the SOC arm as a pre-specified primary analysis of the ITT population. OS is reported here for all participants in the pembro mono arm and SOC arm who were PD-L1 CPS ≥1 (all participants). Per protocol, OS was compared separately between CPS ≥1 participants of the pembro combo arm and SOC arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: All CPS ≥1 participants in the ITT population randomized to the pembro mono arm and SOC arm were analyzed. Per protocol, the pembro combo arm was compared to the SOC arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 256 | 0 | 250
Months | 10.6 [7.7 to 13.8] |  | 11.1 [9.2 to 12.8]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Placebo + SOC Chemotherapy (SOC); OS in CPS ≥1 participants of the pembro mono arm was compared to OS in CPS ≥1 participants of the SOC arm to address the fourth primary hypothesis (non-inferiority to SOC). The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification according to geographic region, disease status, and Fluoropyrimidine treatment; Test type: Non-Inferiority — Pre-specified non-inferiority margin: if the upper bound of the confidence interval (based on the alpha level allocated to the analysis) for the hazard ratio ([HR], pembro mono arm vs SOC) is < 1.2, the pembro mono arm could be considered as non-inferior to the SOC arm in terms of OS; Hazard Ratio (HR) = 0.91, 99.2% CI 2-sided [0.69 to 1.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Placebo + SOC Chemotherapy (SOC); OS in CPS ≥1 participants of the pembro mono arm was compared to OS in CPS ≥1 participants of the SOC arm to address the fifth primary hypothesis (superiority to SOC). The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification according to geographic region, disease status, and Fluoropyrimidine treatment; Test type: Superiority; p = 0.16205, Regression, Cox — One-sided p-value based on log-rank test with stratification; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.74 to 1.10] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Pembro Mono vs SOC: OS in Participants With PD-L1 CPS ≥10
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro mono arm was compared to the SOC arm as a pre-specified primary analysis of the ITT population. OS is reported here for all participants in the pembro mono arm and SOC arm who were PD-L1 CPS ≥10. Per protocol, OS was compared separately between CPS ≥10 participants of the pembro combo arm and SOC arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: All CPS ≥10 participants in the ITT population randomized to the pembro mono arm and SOC arm were analyzed. Per protocol, the pembro combo arm was compared to the SOC arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 92 | 0 | 90
Months | 17.4 [9.1 to 23.1] |  | 10.8 [8.5 to 13.8]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Placebo + SOC Chemotherapy (SOC); OS in CPS ≥10 participants of the pembro mono arm was compared to OS in CPS ≥10 participants of the SOC arm to address the sixth primary hypothesis (superiority to SOC). The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification according to geographic region, disease status, and Fluoropyrimidine treatment; Test type: Superiority; p = 0.01491, Regression, Cox — One-sided p-value based on log-rank test with stratification; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.49 to 0.97] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Pembro Combo vs SOC: Objective Response Rate (ORR) Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1 (All Participants)
Description: ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro combo arm was compared to the SOC arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR for all participants in the pembro combo arm and SOC arm who were PD-L1 CPS ≥1 (all participants). Per protocol, ORR was compared separately between CPS ≥1 participants of the pembro mono arm and SOC arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 0 | 257 | 250
Percentage of Participants |  | 48.6 [42.4 to 54.9] | 37.2 [31.2 to 43.5]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC Chemotherapy (Pembro Combo) vs Placebo + SOC Chemotherapy (SOC); ORR in CPS ≥1 participants of the pembro combo arm was compared to ORR in CPS ≥1 participants of the SOC arm based on Miettinen & Nurminen method stratified by geographic region, disease status, and Fluoropyrimidine treatment; Test type: Other; p = 0.00447, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = 11.5, 95% CI 2-sided [2.9 to 20.0] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Pembro Combo vs SOC: Duration of Response (DOR) Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1 (All Participants)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based upon BICR, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. DOR is reported here for all participants in the pembro combo arm and SOC arm who were PD-L1 CPS ≥1 (all participants) and had CR or PR. Per protocol, DOR was compared separately between CPS ≥1 responders of the pembro mono arm and SOC arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: All CPS ≥1 participants in the ITT population randomized to the pembro combo arm and SOC arm and who demonstrated a confirmed CR or PR were analyzed. Per protocol, the pembro mono arm was compared to the SOC arm separately and not included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 0 | 125 | 93
Months |  | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment) | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment)

8. Secondary Outcome: Pembro Mono vs SOC: ORR Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1 (All Participants)
Description: ORR was defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. Per protocol, ORR in the pembro mono arm was compared to the SOC arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR for all participants in the pembro mono arm and SOC arm who were PD-L1 CPS ≥1 (all participants). Per protocol, ORR was compared separately between CPS ≥1 participants of the pembro combo arm and SOC arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 256 | 0 | 250
Percentage of Participants | 14.8 [10.7 to 19.8] |  | 37.2 [31.2 to 43.5]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Placebo + SOC Chemotherapy (SOC); ORR in CPS ≥1 participants of the pembro mono arm was compared to ORR in CPS ≥1 participants of the SOC arm based on Miettinen & Nurminen method stratified by geographic region, disease status, and Fluoropyrimidine treatment; Test type: Other; p > 0.99999, Miettinen & Nurminen method — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in ORR Percentage = -22.3, 95% CI 2-sided [-29.6 to -14.9] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Pembro Mono vs SOC: DOR Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1 (All Participants)
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based upon BICR, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. DOR is reported here for all participants in the pembro mono arm and SOC arm who were PD-L1 CPS ≥1 (all participants) and had CR or PR. Per protocol, DOR was compared separately between CPS ≥1 responders of the pembro combo arm and SOC arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: All CPS ≥1 participants in the ITT population randomized to the pembro mono arm and SOC arm and who demonstrated a confirmed CR or PR were analyzed. Per protocol, the pembro combo arm was compared to the SOC arm separately and not included in this analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 38 | 0 | 93
Months | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment) |  | NA [NA to NA] — NA=Median DOR and DOR range lower and upper limit not reached (no progressive disease by time of last disease assessment)

10. Secondary Outcome: Pembro Mono vs SOC: PFS Per RECIST 1.1 by BICR in Participants With PD-L1 CPS ≥1 (All Participants)
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
  Per protocol, PFS in the pembro mono arm was compared to the SOC arm as a pre-specified secondary analysis of the ITT population. PFS is reported here for all participants in the pembro mono arm and SOC arm who were PD-L1 CPS ≥1 (all participants). Per protocol, PFS was compared separately between CPS ≥1 participants of the pembro combo arm and SOC arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 256 | 0 | 250
Months | 2.0 [1.5 to 2.8] |  | 6.4 [5.7 to 7.1]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Placebo + SOC Chemotherapy (SOC); PFS in CPS ≥1 participants of the pembro mono arm was compared to PFS in CPS ≥1 participants of the SOC arm based on a Cox regression model with Efron's method of tie handling with treatment as a covariate with stratification according to geographic region, disease status, and fluoropyrimidine treatment; Test type: Other; p = 1.00000, Regression, Cox — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.36 to 1.98] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Pembro Mono vs SOC: Change From Baseline to Week 18 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared between all participants of the pembro mono arm and the SOC arm as a pre-specified secondary analysis. As specified by the protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared separately between all participants of the pembro combo arm and SOC arm and is presented later in the record.
Time Frame: Baseline, Week 18
Population: Participants in the pembro mono arm and SOC arm who received ≥1 dose of study drug and who had EORTC-QLQ-C30 assessments available at baseline or post-baseline up to Week 18. Per protocol, the pembro combo arm was compared to the SOC arm separately and not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 251 | 0 | 243
Score on a Scale | -1.91 [-5.81 to 1.98] |  | -1.75 [-5.17 to 1.66]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Placebo + SOC Chemotherapy (SOC); Change from baseline to Week 18 in EORTC-QLQ-C30 GHS/QoL combined score was compared between all participants of the pembro mono arm and the SOC arm. Comparison based on constrained longitudinal data analysis (cLDA) model with GHS/QoL score as response variable and treatment by visit interaction and stratification factors (geographic region, disease status, and fluoropyrimidine treatment) as covariates; Test type: Other; p = 0.948, cLDA — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in LS Means = -0.16, 95% CI 2-sided [-5.01 to 4.69] — Stratified analyses could be based on collapsing strata with insufficient number of participants or events; strata were pooled in some cases based on clinical judgement and actual counts

12. Secondary Outcome: Pembro Combo vs SOC: Change From Baseline to Week 18 in the EORTC QLQ-C30 Global Health Status/Quality of Life (Items 29 and 30) Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared between all participants of the pembro combo arm and the SOC arm as a pre-specified secondary analysis. As specified by the protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared separately between all participants of the pembro mono arm and SOC arm and is presented earlier in the record.
Time Frame: Baseline, Week 18
Population: Participants in the pembro combo arm and SOC arm who received ≥1 dose of study drug and who had EORTC-QLQ-C30 assessments available at baseline or post-baseline up to Week 18. Per protocol, the pembro mono arm was compared to the SOC arm separately and not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 0 | 245 | 243
Score on a Scale |  | -0.09 [-3.36 to 3.19] | -2.07 [-5.43 to 1.29]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC Chemotherapy (Pembro Combo) vs Placebo + SOC Chemotherapy (SOC); Change from baseline to Week 18 in EORTC-QLQ-C30 GHS/QoL combined score was compared between all participants of the pembro combo arm and the SOC arm. Comparison based on cLDA model with GHS/QoL score as response variable and treatment by visit interaction and stratification factors (geographic region, disease status, and fluoropyrimidine treatment) as covariates; Test type: Other; p = 0.368, cLDA — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in LS Means = 1.98, 95% CI 2-sided [-2.34 to 6.31] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Pembro Mono vs. SOC: Change From Baseline to Week 18 in EORTC QLQ-Module for Gastric Cancer (STO22) Pain Symptom Subscale Score
Description: EORTC-QLQ-STO22 is a 22-item questionnaire developed to assess QoL of gastric cancer participants. It consists of 5 multi-item subscales that assess dysphagia (3 items), dietary restriction (4 items), pain (4 items), upper gastro-esophageal symptoms (3 items), and emotional problems (3 items), and questions on dry mouth, taste, body image, and hair loss. Participant responses to the Pain symptom subscale (Items 34-37) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating more problems. Per protocol, change from baseline to Week 18 in the EORTC-QLQ-STO22 Pain score was compared between the pembro mono arm and the SOC arm as a pre-specified secondary analysis. As specified by the protocol, change from baseline to Week 18 in the EORTC-QLQ-STO22 Pain score was compared separately between the pembro combo arm and SOC arm and is presented later in the record.
Time Frame: Baseline, Week 18
Population: Participants in the pembro mono arm and SOC arm who received ≥1 dose of study drug and who had EORTC-QLQ-STO22 assessments available at baseline or post-baseline up to Week 18. Per protocol, the pembro combo arm was compared to the SOC arm separately and not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 251 | 0 | 243
Score on a Scale | -1.14 [-4.67 to 2.39] |  | -3.49 [-6.60 to -0.38]
Statistical Analysis 1: Comparison: Pembrolizumab Monotherapy (Pembro Mono) vs Placebo + SOC Chemotherapy (SOC); Change from baseline to Week 18 in EORTC-QLQ-STO22 Pain symptom subscale score was compared between all participants of the pembro mono arm and the SOC arm. Comparison based on cLDA model with GHS/QoL score as response variable and treatment by visit interaction and stratification factors (geographic region, disease status, and fluoropyrimidine treatment) as covariates; Test type: Other; p = 0.308, cLDA — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in LS Means = 2.35, 95% CI 2-sided [-2.18 to 6.89] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Pembro Combo vs. SOC: Change From Baseline to Week 18 in EORTC QLQ-STO22 Pain Symptom Subscale Score
Description: EORTC-QLQ-STO22 is a 22-item questionnaire developed to assess QoL of gastric cancer participants. It consists of 5 multi-item subscales that assess dysphagia (3 items), dietary restriction (4 items), pain (4 items), upper gastro-esophageal symptoms (3 items), and emotional problems (3 items), and questions on dry mouth, taste, body image, and hair loss. Participant responses to the Pain symptom subscale (Items 34-37) were scored on a 4-point scale (1=Not at all to 4=Very much). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating more problems. Per protocol, change from baseline to Week 18 in the EORTC-QLQ-STO22 Pain score was compared between the pembro combo arm and the SOC arm as a pre-specified secondary analysis. As specified by the protocol, change from baseline to Week 18 in the EORTC-QLQ-STO22 Pain score was compared separately between the pembro mono arm and SOC arm and is presented earlier in the record.
Time Frame: Baseline, Week 18
Population: Participants in the pembro combo arm and SOC arm who received ≥1 dose of study drug and who had EORTC-QLQ-STO22 assessments available at baseline or post-baseline up to Week 18. Per protocol, the pembro mono arm was compared to the SOC arm separately and not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 0 | 245 | 243
Score on a Scale |  | -10.12 [-13.08 to -7.17] | -3.56 [-6.61 to -0.51]
Statistical Analysis 1: Comparison: Pembrolizumab + SOC Chemotherapy (Pembro Combo) vs Placebo + SOC Chemotherapy (SOC); Change from baseline to Week 18 in EORTC-QLQ-STO22 Pain symptom subscale score was compared between all participants of the pembro combo arm and the SOC arm. Comparison based on cLDA model with GHS/QoL score as response variable and treatment by visit interaction and stratification factors (geographic region, disease status, and fluoropyrimidine treatment) as covariates; Test type: Other; p = 0.001, cLDA — No formal hypothesis testing performed; nominal p-value provided for treatment comparison; Difference in LS Means = -6.56, 95% CI 2-sided [-10.55 to -2.58] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an adverse event. The number of participants who experienced an AE was reported for each arm according to the treatment received.
Time Frame: Up to approximately 33 months
Population: All randomized participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 254 | 250 | 244
Participants | 242 | 244 | 240

16. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an adverse event. The number of participants who discontinued study treatment due to an AE was reported for each arm according to the treatment received.
Time Frame: Up to approximately 30 months
Population: All randomized participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) | Pembrolizumab + SOC Chemotherapy (Pembro Combo) | Placebo + SOC Chemotherapy (SOC)
Number analyzed (Participants) | 254 | 250 | 244
Participants | 29 | 85 | 58

ADVERSE EVENTS:
Time Frame: Up to approximately 78 months
Description: All-Cause Mortality reported for all randomized participants.
  Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab Monotherapy (Pembro Mono) First Course: Participants received pembrolizumab 200 mg IV Q3W.
- Pembrolizumab + SOC Chemotherapy (Pembro Combo)-First Course: Participants received pembrolizumab 200 mg Q3W plus cisplatin 80 mg/m^2 Q3W plus 5-FU 800 mg/m^2/day IV infusion on Days 1-5 Q3W. Capecitabine 1000 mg/m^2 twice a day (BID) on Days 1-14 Q3W could be substituted for 5-FU per local guidelines.
- Placebo + SOC Chemotherapy (SOC)-First Course: Participants received placebo IV Q3W plus cisplatin 80 mg/m^2 Q3W plus 5-FU 800 mg/m^2/day IV infusion on Days 1-5 Q3W. Capecitabine 1000 mg/m^2 BID on Days 1-14 Q3W could be substituted for 5-FU per local guidelines.
- Pembrolizumab Monotherapy Second Course: Eligible participants who stopped the initial course of pembrolizumab (200 mg IV Q3W for up to 35 treatments [approximately 2 years]) with Stable Disease (SD) or better but progressed after discontinuation initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (up to approximately 1 additional year).
- Pembrolizumab + SOC Chemotherapy-Second Course: Eligible participants who stopped the initial course of pembrolizumab (200 mg IV Q3W for up to 35 treatments [approximately 2 years]) administered in combination with SOC chemotherapy, and experienced Stable Disease (SD) or better but progressed after discontinuation initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (up to approximately 1 additional year).
Arm/Group | Pembrolizumab Monotherapy (Pembro Mono) First Course | Pembrolizumab + SOC Chemotherapy (Pembro Combo)-First Course | Placebo + SOC Chemotherapy (SOC)-First Course | Pembrolizumab Monotherapy Second Course | Pembrolizumab + SOC Chemotherapy-Second Course
All-Cause Mortality (participants affected / at risk) | 229/256 | 232/257 | 240/250 | 2/4 | 1/5
Serious Adverse Events (participants affected / at risk) | 93/254 | 122/250 | 117/244 | 1/4 | 0/5
Other Adverse Events (participants affected / at risk) | 216/254 | 239/250 | 234/244 | 3/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy (Pembro Mono) First Course (N=254) | Pembrolizumab + SOC Chemotherapy (Pembro Combo)-First Course (N=250) | Placebo + SOC Chemotherapy (SOC)-First Course (N=244) | Pembrolizumab Monotherapy Second Course (N=4) | Pembrolizumab + SOC Chemotherapy-Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 12 (14) | 10 (13) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 9 (9) | 7 (8) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (7) | 9 (9) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 5 (5) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (7) | 12 (15) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 6 (6) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 5 (5) | 5 (6) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 7 (7) | 8 (10) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 7 (8) | 7 (7) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Refeeding syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 8 (8) | 8 (8) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 13 (13) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy (Pembro Mono) First Course (N=254) | Pembrolizumab + SOC Chemotherapy (Pembro Combo)-First Course (N=250) | Placebo + SOC Chemotherapy (SOC)-First Course (N=244) | Pembrolizumab Monotherapy Second Course (N=4) | Pembrolizumab + SOC Chemotherapy-Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 61 (73) | 112 (150) | 108 (144) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 21 (52) | 26 (51) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 95 (201) | 102 (222) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (5) | 27 (38) | 26 (33) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 22 (24) | 20 (20) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 21 (21) | 28 (29) | 10 (11) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 6 (7) | 2 (2) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 13 (21) | 9 (11) | 10 (10) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 46 (56) | 41 (49) | 41 (54) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 23 (26) | 24 (27) | 23 (25) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 6 (7) | 8 (8) | 14 (15) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 36 (43) | 71 (108) | 68 (83) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 35 (60) | 83 (153) | 71 (106) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 16 (18) | 13 (18) | 11 (13) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 11 (11) | 15 (17) | 16 (20) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 6 (7) | 13 (14) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 49 (59) | 162 (295) | 129 (236) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 33 (49) | 35 (39) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 49 (64) | 84 (148) | 79 (142) | 0 (0) | 0 (0)
Asthenia (General disorders) | 30 (33) | 41 (53) | 47 (81) | 0 (0) | 0 (0)
Chest pain (General disorders) | 4 (6) | 14 (16) | 7 (7) | 0 (0) | 0 (0)
Fatigue (General disorders) | 49 (63) | 105 (156) | 75 (112) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 3 (5) | 41 (57) | 34 (62) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 13 (14) | 16 (16) | 19 (22) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 25 (33) | 32 (38) | 25 (26) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 13 (13) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 13 (16) | 7 (8) | 9 (9) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 18 (22) | 9 (10) | 11 (12) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 8 (8) | 30 (52) | 34 (59) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (15) | 59 (120) | 40 (79) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 23 (38) | 17 (21) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 28 (28) | 54 (63) | 33 (33) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 4 (6) | 30 (71) | 25 (52) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 48 (53) | 94 (135) | 90 (127) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 11 (14) | 16 (19) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 (21) | 17 (21) | 23 (28) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (10) | 14 (20) | 14 (16) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (16) | 35 (49) | 42 (61) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (11) | 34 (43) | 32 (48) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (16) | 12 (21) | 20 (26) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 15 (21) | 9 (16) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (20) | 22 (25) | 7 (7) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (32) | 13 (14) | 14 (15) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 17 (23) | 8 (9) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 14 (18) | 20 (21) | 15 (22) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 16 (18) | 20 (21) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (18) | 24 (26) | 16 (22) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 31 (36) | 16 (17) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 34 (37) | 16 (18) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 21 (21) | 18 (19) | 22 (24) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 24 (26) | 23 (26) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 19 (23) | 9 (11) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 10 (12) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 16 (20) | 12 (21) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 19 (19) | 11 (11) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 15 (16) | 15 (15) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 60 (69) | 46 (57) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (27) | 21 (25) | 8 (11) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 20 (23) | 31 (41) | 15 (18) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 11 (12) | 10 (13) | 12 (17) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT02494583/Prot_SAP_000.pdf